CLINICAL TRIAL: NCT00030550
Title: A Randomized, Multi-Center, Double-Blind, Placebo-Controlled Trial Assessing The Safety And Efficacy Of Thalidomide (THALOMID) For The Treatment Of Anemia In Red Blood Cell Transfusion-Dependent Patients With Myelodysplastic Syndromes
Brief Title: Thalidomide in Treating Anemia in Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: DS 01-16; RPCI-DS-0116; CELGENE-T-MDS-001; NCI-G01-2044
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; de novo myelodysplastic syndromes; chronic myelomonocytic leukemia; previously treated myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; atypical chronic myeloid leukemia, BCR-ABL1 negative
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may be an effective treatment for anemia caused by myelodysplastic syndrome.

PURPOSE: Randomized phase II trial to study the effectiveness of thalidomide in treating anemia in patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of thalidomide for the treatment of anemia in patients with myelodysplastic syndromes.
* Determine whether this drug reduces the frequency of leukemia transformation and decreases bone marrow blast percentage in these patients.
* Determine the effect of this drug on neutrophil and platelet production and the number of episodes of febrile neutropenia in these patients.
* Determine the safety of this drug in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to International Prognostic Scoring System score (low and intermediate-1 vs intermediate-2 and high) and transfusion dependence (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oral thalidomide once daily on weeks 1-24.
* Arm II: Patients receive oral placebo once daily on weeks 1-24. In both arms, patients who have not progressed to leukemia after 24 weeks of therapy may receive open-label thalidomide for an additional 24 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 220 patients (110 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelodysplastic syndromes (MDS) of at least 12 weeks duration

  * Refractory anemia (RA)
  * RA with ringed sideroblasts
  * RA with excess blasts
  * Chronic myelomonocytic
* No therapy-related MDS
* No myelosclerosis or myelofibrosis occupying more than 30% of marrow space (or assessed as grade 3+ or greater)
* No transformation to acute myeloid leukemia
* No more than 20% blasts in bone marrow
* No more than 5% blasts in peripheral blood
* Patients with an erythropoietin level 100 mU/mL or less must have failed epoetin alfa treatment (i.e., at least 30,000 units of epoetin alfa weekly for at least 6 weeks)
* Transfusion-dependent (received at least 2 units of packed RBCs or whole blood within the past 8 weeks) OR
* Transfusion-independent (no packed RBC or whole blood transfusions within the past 8 weeks with 2 hemoglobin levels (at least 7 days apart) less than 11 g/dL)
* No iron deficiency (e.g., absent bone marrow iron store)

  * If marrow aspirate is not evaluable, transferrin saturation must be at least 20% and ferritin at least 50 ng/mL
* No uncorrected B12 or folate deficiency
* No other contributing causes of anemia (e.g., autoimmune or hereditary hemolytic disorders or gastrointestinal blood loss)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Zubrod 0-2

Life expectancy:

* At least 6 months

Hematopoietic:

* See Disease Characteristics
* Absolute neutrophil count at least 500/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST and ALT less than 2 times upper limit of normal (ULN)
* Hepatitis B surface antigen negative
* Hepatitis C negative

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No uncontrolled hypertension
* No clinically significant, symptomatic, unstable cardiovascular disease unrelated to MDS

Pulmonary:

* No clinically significant, symptomatic, unstable pulmonary disease unrelated to MDS

Neurologic:

* No clinically significant, symptomatic, unstable neurologic disease unrelated to MDS
* No history of epilepsy
* No sustained neurologic deficit (e.g., stroke)
* No grade 2 or greater peripheral neuropathy

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use at least 1 highly effective and 1 additional effective method of contraception for 4 weeks prior to, during, and for 4 weeks after study participation
* HIV negative
* No clinically significant, symptomatic, unstable endocrine, gastrointestinal, or genitourinary disease unrelated to MDS
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No life-threatening or active infection requiring parenteral antibiotics
* No other serious concurrent illness

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* More than 7 days since prior hematopoietic growth factors (e.g., epoetin alfa, filgrastim (G-CSF), sargramostim (GM-CSF), or interleukin-3)
* No prior thalidomide
* No prior agents intended to inhibit vascular endothelial growth factor or tumor necrosis factor alfa (e.g., etanercept or infliximab)
* No concurrent epoetin alfa

Chemotherapy:

* No concurrent chemotherapy that may be active against MDS

Endocrine therapy:

* More than 30 days since prior androgens
* No requirement for ongoing therapy with systemic corticosteroids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* More than 30 days since prior treatment for MDS except RBC transfusion or epoetin alfa
* More than 30 days since prior participation in another experimental clinical trial
* More than 30 days since prior experimental drugs
* No other concurrent investigational agents or treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L. Slack, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- PPD Development, Wilmington, North Carolina, United States